CLINICAL TRIAL: NCT01246856
Title: MIBG Scintigraphy and Strain Echocardiography in the Detection of Subclinical Cardiovascular Effects One Year After (Neo)Adjuvant Breast Cancer Treatment With Docetaxel, Doxorubicin and Cyclophosphamide (TAC)
Brief Title: MIBG Scintigraphy and Strain Echocardiography in the Detection of Subclinical Cardiovascular Effects One Year After (Neo)Adjuvant Breast Cancer Treatment With Docetaxel, Doxorubicin and Cyclophosphamide (TAC): a Pilot Study
Acronym: TOXTAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCNONCO201005
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Breast Cancer
Keywords: Cardiotoxicity; Breast cancer treatment; MIBG scintigraphy; Strain Echocardiography; patients who have been treated with TAC one year previously
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
Many patients with breastcancer in the past, were treated with TAC. These last years, there is more and more focus on the effects of chemotherapy, particularly in children treated with this. One of these effects is damage to the heart muscle, which ultimately might affect the pump-function of the heart . In adults, the effect of treatment with TAC on the heart, has not been previously investigated. The possibility exists that the adverse reactions in children are found in adults also could occur. Therefore we have initiated this trial.

DETAILED DESCRIPTION:
Given the lack of data on the incidence of subclinical cardiotoxicity after treatment with TAC we want to assess whether subclinical cardiovascular damage is present in adult patients with breast cancer who have completed treatment with (neo)adjuvant TAC one year previously, using MIBG (meta-iodobenzylguanidine) scintigraphy, novel echocardiographic techniques and blood biomarkers. Following the study by Lipshultz et al. we expect to find at least in 25% of the patients signs of subclinical cardiovascular damage with at least one of the three techniques.(11) If at least 10% is observed we will conclude that it is useful to further pursue the use of these techniques for the detection of subclinical cardiotoxicity in a next clinical study which will be powered to assess the predictive value of these techniques for the development of clinical heart failure. If a lower percentage is observed we will conclude that it is not useful to further pursue the use of these techniques for the detection of subclinical cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer, ≥ 18 years old at the time of breast cancer diagnosis
* (Neo)adjuvant treatment with docetaxel, doxorubicin and cyclophosphamide (TAC) completed one year before inclusion

Exclusion Criteria:

* Evidence of breast cancer recurrence or metastatic disease
* Evidence of heart disease at the time of breast cancer diagnosis
* Evidence of renal failure at the time of cardiac evaluation
* Pregnant or lactating
* Participation in a research protocol with ionizing radiation within one year before inclusion.
* Evidence of diabetes mellitus or Parkinson's disease
* Evidence of an MIBG-accumulating tumor (pheochromocytoma, paraganglioma, chemodectoma, ganglioneuroma, neuroblastoma, carcinoid, medullary thyroid cancer, neurofibromatosis, retinoblastoma, esthesioneuroma, schwannoma, merkelcel-tumor, pancreatic islet cell tumors, small cell lung carcinoma, melanoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been treated with TAC one year previously
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: H.W.M. van Laarhoven, Md, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands